CLINICAL TRIAL: NCT05595811
Title: The Outcome After Operation for Pancreatic and Periampullary Tumors in Greeland Inuit.
Brief Title: Pancreatic and Periampullary Tumors in Greenland Inuit
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, carsten palnaes hansen, consultant, Rigshospitalet, Denmark
Other Study IDs: RH-C-2022-1
Record Dates: First submitted 2022-10-14; First posted 2022-10-27 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Neoplasms; Periampullary Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inuit: Inuit living in Greenland
  Interventions: Other: outcome following surgery
- Danish: Danish patients living in Denmark
  Interventions: Other: outcome following surgery

INTERVENTIONS:
Other: outcome following surgery

SUMMARY:
Especially since the Second World War the indigenous population in the Arctic, the Inuit have gone through a Westernization, which has improved the health conditions but also changed the disease panorama with an increasing incidence of cancer. This is exemplified by a decrease in physical activity, due to the depletion of the Greenlandic hunting traditions, tobacco smoking and unhealthy diet. At the beginning of the westernization, malignant diseases were highly uncommon, but they started to increase due to the increasing life expectancy and changes in lifestyle. The incidence of pancreatic and periampullary cancer has been reported to be the same among Inuit in Canada, Denmark, and the United States but with a higher incidence than among the Caucasian population in the three countries.

The aim with this study was to investigate the results of pancreatic surgery for pancreatic and periampullary tumors in Inuit patients in Greenland at to compare the outcome of surgery and the overall survival with a cohort of Danish patients.

DETAILED DESCRIPTION:
Study design. The study is a retrospective, descriptive register study based on data from a prospectively maintained database. The study is a comparison of two cohorts, all Inuit patients living in Greenland, who had pancreatic operations for pancreatic and periampullary tumors - either preoperatively verified or suspected - at Rigshospitalet, Copenhagen University Hospital from 31. January 1999 to 31. January 2021. Danish patients living in Greenland were not included in the study. Inuit patients were compared with a cohort of Danish patients with same diagnosis and same range of age operated during the same period at the hospital. All diagnoses were histologically verified. Data recruitment include all patients operated between January 31, 1999 and January 31, 2021 with follow-up until December 31 after which data will be evaluated. The study is reported according to the STROCSS guidelines (www.strocssguideline.com).

Study population. The study includes 2326 consecutive patients, 47 inuit and 2279 Danish patients between 41 and 79 years (age range based on the inuit patients). There are 1,208 patients with malignant tumours of whom 1,020 have adenocarcinoma.

Data collection Data are collected from our prospectively maintained database of pancreatic operations, from the electronic hospital record systems Orbit and EPIC, the Danish National Pathology Data Registry, and from the National Register of Death. All Danish Nationals including citizens in Greenland have a unique Central Person Registration number that enables searching of health data.

Outcomes. Relevant postoperative complications are recorded in the study and include leakage from the pancreatic, bile or gastrojejunal anastomosis, intraabdominal hemorrhage and abscess formation or other complications with severe or fatal outcome. Outcomes are defined as postoperative complications and mortality assessed during 30- and 90-days and overall survival (OS) defined as the time from surgery to death from any cause or censoring at time of last follow-up. Hospitalization is defined as postoperative stay until discharge. In-hospital mortality is defined as all deaths from time of admission until discharge. Cancer specific mortality is defined as death from adenocarcinoma after other causes are censured.

Statistics. Data are presented as median and range if not otherwise stated. Categorial data are presented as numbers or percentage and are analyzed with Fisher's exact test. Non-parametric continuous data between subgroups are analyzed with the Mann-Whitney test. The Kaplan-Meier method and the cumulative incidence function with correction for competing risks are used to estimate OS and the log-rank test to examine the differences between curves. The reference population is an age and sex matched Danish standard population. A p < 0.05 is considered statistically significant. Statistical analysis is performed with GraphPad Prism software version 6.05. (GraphPad, La Jolla, CA).

Ethics. The study is a descriptive study and conducted in accordance with the principles stated in the Declaration of Helsinki. No approval is required according to the Danish National Health Board. The study is an observational, retrospective quality assurance project according to the guidelines of the Danish Health Data Authority (http://Sundhedsdatastyrelsen.dk). No approval is required according to the Danish National Health Board. In this respect it has to be noticed that a major part of the Greenlandic and Danish patients had died before the study was initiated, and the Regional Ethical Committee of the Capital Region of Denmark provided exemption for the study. The use of register data follows the General Data Protection Regulation of the European Union and the Danish Data Protection Agency. Patients' written consent for using health data was obtained before operation. The study and the use of data were consented by the hospital ethical

ELIGIBILITY:
Inclusion Criteria:

* Greenland Inuit patients
* operated for pancreatic and periampullary cancer
* time of operation 31. January 1999 to 31. January 2021
* sex: all
* minimum age: 41 years
* maximum years: 79 years

Exclusion Criteria

* patients beyond the age limit
* patients operated beyond the time limit

Danish patients

* operated for pancreatic and periampullary cancer
* time of operation 31. January 1999 to 31. January 2021
* sex: all
* minimum age: 41 years
* maximum years: 79 years

Exclusion Criteria: patients beyond the age limit.

* patients beyond the age limit.
* time of operation 31. January 1999 to 31. January 2021

Ages: 41 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Greenland Inuit, both sex, living in Greenland and operated at Copenhagen University Hospital Rigshospitalet Danish patients (controls), both sex living in Denmark and operated at Copenhagen University Hospital Rigshospitalet
Sampling Method: Non-Probability Sample
Enrollment: 2326 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
waiting time from diagnosis to surgery | from 31. January 1999 to 31. January 2021
  time from diagnosis to surgery for each patient
number and kind of postoperative complications | 31. January 1999 to 31. January 2021
  anastomosis leak, bleeding, death of any reason, in-hospital
overall survival | 31. January 1999 to 31. January 2022
  from operation to death of any course

SECONDARY OUTCOMES:
adjuvant oncologic treatment | 31. January 1999 to 31. January 2021
  numbers treated

CONTACTS AND LOCATIONS:
Overall Officials: carsten p hansen, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] GBD 2017 Pancreatic Cancer Collaborators. The global, regional, and national burden of pancreatic cancer and its attributable risk factors in 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Gastroenterol Hepatol. 2019 Dec;4(12):934-947. doi: 10.1016/S2468-1253(19)30347-4. Epub 2019 Oct 21. PMID 31648972
- [Background] Rawla P, Sunkara T, Gaduputi V. Epidemiology of Pancreatic Cancer: Global Trends, Etiology and Risk Factors. World J Oncol. 2019 Feb;10(1):10-27. doi: 10.14740/wjon1166. Epub 2019 Feb 26. PMID 30834048
- [Background] Bjerregaard P, Curtis T, Borch-Johnsen K, Mulvad G, Becker U, Andersen S, Backer V. Inuit health in Greenland: a population survey of life style and disease in Greenland and among Inuit living in Denmark. Int J Circumpolar Health. 2003;62 Suppl 1:3-79. doi: 10.3402/ijch.v62i0.18212. PMID 14527126
- [Background] Friborg JT, Melbye M. Cancer patterns in Inuit populations. Lancet Oncol. 2008 Sep;9(9):892-900. doi: 10.1016/S1470-2045(08)70231-6. PMID 18760245
- [Background] Circumpolar Inuit Cancer Review Working Group; Kelly J, Lanier A, Santos M, Healey S, Louchini R, Friborg J, Young K, Ng C. Cancer among the circumpolar Inuit, 1989-2003. I. Background and methods. Int J Circumpolar Health. 2008 Dec;67(5):396-407. doi: 10.3402/ijch.v67i5.18348. PMID 19186761
- [Background] Yousaf U, Engholm G, Storm H, Christensen N, Zetlitz E, Trykker H, Sejersen F, Bjerregaard P, Thygesen LC. Cancer Incidence and Mortality in Greenland 1983-2014 - Including Comparison With the Other Nordic Countries. EClinicalMedicine. 2018 Aug 29;2-3:37-49. doi: 10.1016/j.eclinm.2018.08.003. eCollection 2018 Aug-Sep. PMID 31193566
- [Background] Schmidt M, Pedersen L, Sorensen HT. The Danish Civil Registration System as a tool in epidemiology. Eur J Epidemiol. 2014 Aug;29(8):541-9. doi: 10.1007/s10654-014-9930-3. Epub 2014 Jun 26. PMID 24965263
- [Background] Valle JW, Palmer D, Jackson R, Cox T, Neoptolemos JP, Ghaneh P, Rawcliffe CL, Bassi C, Stocken DD, Cunningham D, O'Reilly D, Goldstein D, Robinson BA, Karapetis C, Scarfe A, Lacaine F, Sand J, Izbicki JR, Mayerle J, Dervenis C, Olah A, Butturini G, Lind PA, Middleton MR, Anthoney A, Sumpter K, Carter R, Buchler MW. Optimal duration and timing of adjuvant chemotherapy after definitive surgery for ductal adenocarcinoma of the pancreas: ongoing lessons from the ESPAC-3 study. J Clin Oncol. 2014 Feb 20;32(6):504-12. doi: 10.1200/JCO.2013.50.7657. Epub 2014 Jan 13. PMID 24419109
- [Background] Neoptolemos JP, Palmer DH, Ghaneh P, Psarelli EE, Valle JW, Halloran CM, Faluyi O, O'Reilly DA, Cunningham D, Wadsley J, Darby S, Meyer T, Gillmore R, Anthoney A, Lind P, Glimelius B, Falk S, Izbicki JR, Middleton GW, Cummins S, Ross PJ, Wasan H, McDonald A, Crosby T, Ma YT, Patel K, Sherriff D, Soomal R, Borg D, Sothi S, Hammel P, Hackert T, Jackson R, Buchler MW; European Study Group for Pancreatic Cancer. Comparison of adjuvant gemcitabine and capecitabine with gemcitabine monotherapy in patients with resected pancreatic cancer (ESPAC-4): a multicentre, open-label, randomised, phase 3 trial. Lancet. 2017 Mar 11;389(10073):1011-1024. doi: 10.1016/S0140-6736(16)32409-6. Epub 2017 Jan 25. PMID 28129987
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Mathew G, Agha R; STROCSS Group. STROCSS 2021: Strengthening the reporting of cohort, cross-sectional and case-control studies in surgery. Ann Med Surg (Lond). 2021 Nov 6;72:103026. doi: 10.1016/j.amsu.2021.103026. eCollection 2021 Dec. PMID 34820121
- [Background] Storm HH, Nielsen NH. Cancer of the digestive system in Circumpolar Inuit. Acta Oncol. 1996;35(5):553-70. doi: 10.3109/02841869609096987. PMID 8813062
- [Background] Kirkegaard J. Incidence of pancreatic cancer in Greenland 2000-2010. Int J Circumpolar Health. 2012 May 22;71:18368. doi: 10.3402/ijch.v71i0.18368. PMID 22663941
- [Background] Young TK, Kelly JJ, Friborg J, Soininen L, Wong KO. Cancer among circumpolar populations: an emerging public health concern. Int J Circumpolar Health. 2016 Jan 12;75:29787. doi: 10.3402/ijch.v75.29787. eCollection 2016. PMID 26765259
- [Background] Alberts SR, Kelly JJ, Ashokkumar R, Lanier AP. Occurrence of pancreatic, biliary tract, and gallbladder cancers in Alaska Native people, 1973-2007. Int J Circumpolar Health. 2012 Mar 20;71:17521. doi: 10.3402/IJCH.v71i0.17521. PMID 22456038
- [Background] Engholm G, Ferlay J, Christensen N, Bray F, Gjerstorff ML, Klint A, Kotlum JE, Olafsdottir E, Pukkala E, Storm HH. NORDCAN--a Nordic tool for cancer information, planning, quality control and research. Acta Oncol. 2010 Jun;49(5):725-36. doi: 10.3109/02841861003782017. PMID 20491528
- [Background] Bosetti C, Lucenteforte E, Silverman DT, Petersen G, Bracci PM, Ji BT, Negri E, Li D, Risch HA, Olson SH, Gallinger S, Miller AB, Bueno-de-Mesquita HB, Talamini R, Polesel J, Ghadirian P, Baghurst PA, Zatonski W, Fontham E, Bamlet WR, Holly EA, Bertuccio P, Gao YT, Hassan M, Yu H, Kurtz RC, Cotterchio M, Su J, Maisonneuve P, Duell EJ, Boffetta P, La Vecchia C. Cigarette smoking and pancreatic cancer: an analysis from the International Pancreatic Cancer Case-Control Consortium (Panc4). Ann Oncol. 2012 Jul;23(7):1880-8. doi: 10.1093/annonc/mdr541. Epub 2011 Nov 21. PMID 22104574
- [Background] Weissman S, Takakura K, Eibl G, Pandol SJ, Saruta M. The Diverse Involvement of Cigarette Smoking in Pancreatic Cancer Development and Prognosis. Pancreas. 2020 May/Jun;49(5):612-620. doi: 10.1097/MPA.0000000000001550. PMID 32433397
- [Background] Senftleber NK, Overvad M, Dahl-Petersen IK, Bjerregaard P, Jorgensen ME. Diet and physical activity in Greenland: genetic interactions and associations with obesity and diabetes. Appl Physiol Nutr Metab. 2021 Aug;46(8):849-855. doi: 10.1139/apnm-2021-0020. Epub 2021 Jun 9. PMID 34107227
- [Background] Bjerregaard P, Larsen CVL. Social determinants of dietary patterns, food basket costs and expenditure on alcohol and tobacco amongst Greenland Inuit. Public Health Nutr. 2021 Oct;24(15):4975-4984. doi: 10.1017/S1368980020005133. Epub 2021 Jan 19. PMID 33461645
- [Background] Pedersen ML. Diabetes mellitus in Greenland. Dan Med J. 2012 Feb;59(2):B4386. PMID 22293056
- [Background] Carstensen B, Ronn PF, Jorgensen ME. Prevalence, incidence and mortality of type 1 and type 2 diabetes in Denmark 1996-2016. BMJ Open Diabetes Res Care. 2020 May;8(1):e001071. doi: 10.1136/bmjdrc-2019-001071. PMID 32475839
- [Background] Nielsen MH, Backe MB, Pedersen ML. Prevalence of patients using antihypertensive medication in Greenland, and an assessment of the importance of diagnosis for the associated quality of care - a cross-sectional study. Int J Circumpolar Health. 2022 Dec;81(1):2110675. doi: 10.1080/22423982.2022.2110675. PMID 35938701
- [Background] Lavoie JG, Stoor JP, Rink E, Cueva K, Gladun E, Larsen CVL, Healey Akearok G, Kanayurak N. Cultural competence and safety in Circumpolar countries: an analysis of discourses in healthcare. Int J Circumpolar Health. 2022 Dec;81(1):2055728. doi: 10.1080/22423982.2022.2055728. PMID 35451927
- [Background] Tolstrup J, Madsen RC, Sneftrup MV, Niclasen B. Greenlandic patients with colorectal cancer: symptomatology, primary investigations and differences in diagnostic intervals between Nuuk and the rest of the country. Int J Circumpolar Health. 2017;76(1):1344086. doi: 10.1080/22423982.2017.1344086. PMID 28705121
- [Background] van Walraven C, McAlister FA. Competing risk bias was common in Kaplan-Meier risk estimates published in prominent medical journals. J Clin Epidemiol. 2016 Jan;69:170-3.e8. doi: 10.1016/j.jclinepi.2015.07.006. Epub 2015 Jul 29. PMID 26232083
- [Background] Augustussen M, Hounsgaard L, Pedersen ML, Sjogren P, Timm H. Relatives' level of satisfaction with advanced cancer care in Greenland - a mixed methods study. Int J Circumpolar Health. 2017;76(1):1335148. doi: 10.1080/22423982.2017.1335148. PMID 28613119